CLINICAL TRIAL: NCT05868629
Title: Clinical Study To Further Evaluate The Efficacy Of Dabrafenib Plus Trametinib In Patients With Rare BRAF V600E Mutation-Positive Unresectable or Metastatic Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CDRB436IIC01
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Rare Unresectable or Metastatic BRAF V600E Mutation-positive Solid Tumors
Keywords: BRAF; v-raf murine sarcoma viral oncogene homolog B1; dabrafenib; trametinib; tumor agnostic
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- dabrafenib plus trametinib: patients treated with dabrafenib and trametinib
  Interventions: Other: Non-investigational

INTERVENTIONS:
Other: Non-investigational — Participants obtaining commercial (non-investigational) dabrafenib plus trametinib (i.e. solid formulation or liquid formulation, if approved and commercially available locally) per local guidance or patient access program

SUMMARY:
This study is a phase IV, pragmatic single-arm prospective, open label study in pediatric (1 years or older) and adult study participants with rare BRAF V600E mutation-positive unresectable or metastatic solid tumors for whom a decision has already been made to be treated with dabrafenib and trametinib, irrespective of the trial participation.

ELIGIBILITY:
Inclusion Criteria:

* Study participant with a BRAF V600E mutation-positive solid tumor as confirmed by a local laboratory test;
* At least 1 measurable lesion as defined by RECIST v1.1 per local review;
* Study participant previously not treated with dabrafenib and/or trametinib. Study participants who received dabrafenib and trametinib in the past for the treatment of other malignancies are eligible if treatment has been discontinued for greater than 1 year;
* Ability to provide scans for central imaging review

Exclusion Criteria:

* Those with the following tumor types: melanoma, NSCLC, ATC, BTC, glioma and CRC;
* Study participants who have contraindication to receive dabrafenib and/ or trametinib according to the local label;

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants diagnosed with a rare BRAF V600E mutation-positive unresectable or metastatic solid tumor, 1 year and older excluding patients with melanoma, Non-Small Cell Lung Cancer, Colorectal Cancer, Anaplastic Thyroid Cancer, Biliary Tract Cancer and glioma, who will be treated with dabrafenib and trametinib.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2028-03-03 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 4 years
  Proportion of study participants with a best overall confirmed Complete Response (CR) or Partial Response (PR) by independent central review according to RECIST v1.1 or other relevant response criteria.

SECONDARY OUTCOMES:
Duration of response (DOR) | Approximately 4 years
  Defined as time from the onset of tumor response until the date of the first documented progressive disease (PD) or death due to any cause.
Clinical benefit rate (CBR) | Approximately 4 years
  Defined as the proportion of study participants with a best overall response of CR, PR or stable disease (SD), lasting as per independent central review, for a duration of at least 24 weeks. CR, PR and SD are defined according to RECIST v1.1. or other relevant response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (7):
  - Lundquist Inst BioMed at Harbor, Torrance, California
  - Johns Hopkins University, Washington D.C., District of Columbia
  - Duke Clinical Research Institute, Durham, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - El Paso Texas Oncology, El Paso, Texas
  - Texas Oncology San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No